CLINICAL TRIAL: NCT01422252
Title: Evaluation of Falls Occurring at Home in People Over 75 Equipped or Non-equipped With a Precocious Detection Device. Prospective Interventional Study.
Brief Title: Evaluation of a Fall Detection Device in Isolated Elderly
Acronym: VIGI91
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more inclusions
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vigilio S.A. (Unknown); Hôpital Privé Gériatrique Les Magnolias (HPGM) (Unknown); Conseil Général de l'Essonne (Unknown); SDIS de l'Essonne (Unknown); SAMU de l'Essonne (Unknown); Europ Assistance (Unknown); Réseau Hippocampes (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P100202
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Accidental Falls; Elderly
Keywords: Falls Elderly persons; Isolated At risk for falls; Fall detection device; Precocious detection Vigi'Fall®

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Persons equipped (Experimental): Precocious fall detection device
  Interventions: Device: Vigi'Fall®
- Persons non-equipped (No Intervention): No fall detection device

INTERVENTIONS:
Device: Vigi'Fall® — Precocious fall detection device
  Arms: Persons equipped

SUMMARY:
The objective of this study is to evaluate the evolution 6 months after a fall occurring at home in people over 75 equipped or non-equipped with a precocious detection device. The possibility to establish a relation between the alert emitted by the device, the time separating the fall from the arrival at hospital and the potential consequences for the persons will be analyzed with the greatest accuracy. Besides, the sequences of intervention of the different operators will be described with precision. 200 persons living at home in the ESSONNE(France)and having fallen at least one time during the previous 3 months will be included in the study and two groups of 100 will be constituted randomly after having signed a written consent. Of the 2 groups, one will be constituted with persons equipped with a precocious fall detection device named Vigi'Fall® , the second being non-equipped. After a first visit checking that the inclusion criteria are abide by and the installation of the device in the persons designated randomly for being equipped, a second visit will be carried out after 10 months in order to know the evolution, i.e. if the persons are still alive, living at home or having left for admission in an institution (hospital, nursing home, retirement home...). By a detailed comparison between the 2 groups, it will be possible to evaluate the potential interest of having been equipped or non-equipped with a precocious fall detection device. Hence, a change in practices may lead to a prevision of elderly persons likely to benefit of a precocious detection device and to the development of prevention in hospital geriatric departments, geriatric care networks, emergency departments and local services for the elderly and disabled. Another possible gain of the study is to sensitize the medical, paramedical and social teams to the usefulness of precocious detection devices in elderly subjects at risk for falls.

DETAILED DESCRIPTION:
Objectives of the study:

Principal objective : To evaluate the evolution 6 months after a fall occurring at home in people over 75 equipped or non-equipped with a precocious detection device. Prospective interventional study.

Secondary objective : To establish a relation between the alert emitted by the device, the time separating the fall from the arrival at hospital and the potential MORBI-mortality To describe the sequences of intervention of the different operators Methodology :Multicenter, prospective, cohort, interventional study. Pattern of the study : The study will comprehend 2 visits to be realized in a 10-month interval.

Visits:

1. Randomization, inclusion and selection visit(Visit 1): The inclusion of the subject will be effective once the enlightened consent signed, after check of the inclusion criteria. Inclusion and standardized questioning will be realized by the medical evaluators. The data will be obtained by questioning the subject and if need be of relatives and GP. The questioning will be carried out with a questionnaire on independent card comprising the frailty elements. Independently, a follow-up will be operated at home by a nurse of HPGM Les Magnolias hospital for the maintenance of the adhesive patch to be changed regularly nearly every 10 days in the persons equipped, the study plans the installation of Vigi'Fall® device as the only peculiar measure during the coverage. At the conclusion of that first report, the whole questionnaires will be picked up again by a participant in charge of completing the potential missing data. Via this colligation of missing data, the exhaustiveness of the data will be automatically checked.
2. End of study visit (Visit 2): 10 months 10 months after the installation of Vigi'Fall® device, a contact will be established with the subject and if need be relatives and GP to be informed of the evolution but as well the appearance of potential falls with their characteristics.

   * Relation between alert, intervention time and evolution : Theses relations will be investigated with the most possible accuracy. The standardized questioning will be completed by an investigator up to a maximal exhaustiveness.
   * Description of the sequences of intervention:These sequences will be evaluated via a simple and standardized questionnaire.
   * Expected results, perspectives and scientific data: To quantify with accuracy the evolution in persons over 75 equipped with a precocious detection device after a fall occurring at home in comparison with a witness population non equipped. To establish a relation between the alert emitted by the device, the time separating the fall from the arrival at hospital and the potential MORBI-mortality. To describe with the most possible accuracy the time sequences of the different operators To quantify the rate of subjects hospitalized (with the duration of hospitalization), of subjects still living at home or having left to be admitted in institution (nursing home, retirement home...) in the different groups. The information hence obtained will enable a better knowledge of the tools for detection and precocious alert in falls of the elderly.
   * Direct benefit for geriatricians, sanitary and care professionals and emergency physicians:

Change in practices :Prevision of subjects likely to benefit of a precocious detection device. Development of prevention in hospital geriatric departments, geriatric care networks, emergency departments and local services for the elderly and disabled (SDPAH).

Education : Sensitize the medical, paramedical and social teams to the usefulness of precocious detection devices in elderly subjects at risk for falls.

ELIGIBILITY:
Inclusion Criteria:

* Person over 75 living at home alone in ESSONNE (France) and having fallen at least one time during the 3 months preceding the inclusion in the study.
* Person having signed a free and enlightened consent

Exclusion Criteria:

* Person living in institution (nursing home, retirement home...)
* Person under 75
* Person with severe cognitive impairment (MMS < 15)
* Person under protection as incapable (guardianship or trusteeship)
* Person not affiliated to a social insurance

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Death | 6 months
  The death 6 months after a recurrent fall

SECONDARY OUTCOMES:
Time between the fall and the arrival of emergency | 13 months
  The time between the fall and the arrival of emergency will be compared in both groups.
Hospitalization | 13 months
  The rate of subjects hospitalized (with the duration of hospitalization)
Follow up of patients | 13 months
  The rate of subjects still living at home or having left to be admitted in an institution (nursing home, retirement home...).

CONTACTS AND LOCATIONS:
Overall Officials: Yann-Erick Claessens, MD, PhD, Principal Investigator — Hôpital Cochin
Locations (1):
- Cochin Hospital, Paris, France